CLINICAL TRIAL: NCT01340989
Title: Evaluation of Adding 4% of Oxygen and 10% of Nitrous Oxide to the CO2 Pneumoperitoneum Upon CO2 Resorption.
Brief Title: CO2 Absorption During Laparoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Gasthuisberg (Other)
Responsible Party: Principal Investigator, Jasper Verguts, MD, University Hospital, Gasthuisberg
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: s52645
Record Dates: First submitted 2011-04-21; First posted 2011-04-25 (Estimated); Last update posted 2011-10-26 (Estimated); Status verified 2011-10

CONDITIONS: Pneumoperitoneum
Keywords: women undergoing laparoscopic surgery for: hysterectomy, colpopexy, endometriosis, adhesions or myomas
MeSH Terms: conditions — Pneumoperitoneum; Endometriosis; Tissue Adhesions; Myoma

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- 4% oxygen (Experimental): addition of 4% oxygen to the CO2 pneumoperitoneum
  Interventions: Procedure: alteration of the insufflation gas
- full conditioning (Experimental): full conditioning of the peritoneal cavity by the laparoscopic gas: 4% oxygen, 10% nitrous oxide, humidification and set temperature of 32°C
  Interventions: Procedure: full conditioning
- CO2 pneumoperitoneum (Active Comparator): standard laparoscopy with CO2 pneumoperitoneum
  Interventions: Procedure: standard pneumoperitoneum

INTERVENTIONS:
Procedure: alteration of the insufflation gas — addition of 4% oxygen
  Arms: 4% oxygen
Procedure: full conditioning — addition of 4% oxygen + 10% nitrous oxide to the peritoneum
  * humidification
  * set temperature of 32°C
  Arms: full conditioning
Procedure: standard pneumoperitoneum — no intervention besides the use of CO2
  Arms: CO2 pneumoperitoneum

SUMMARY:
CO2 absorption from the pneumoperitoneum increases over time during laparoscopic procedures. Adding 4% of oxygen to the carbon dioxide was shown in rabbits to decrease CO2 resorbtion through prevention of mesothelial hypoxia. We want to prove this concept in human and expand it to the use of full conditioning.

DETAILED DESCRIPTION:
In order to confirm the animal data in the human, a first RCT was performed in which 20 women undergoing a laparoscopy for at least 60 minutes were randomised to a pneumoperitoneum with either 100% carbon dioxide or 96% carbon dioxide plus 4% of oxygen. Insufflation pressure and Trendelenburg were standardised at 15 mm Hg and 30° respectively. In a second trial women were randomized to either 100% carbon dioxide or 86% carbon dioxide plus 4% of oxygen + 10% nitrous oxide + humidification and set temperature of 32°C of the peritoneal cavity.

ELIGIBILITY:
Inclusion Criteria:

* Women/men planned to undergo a laparoscopic intervention for at least 1 hour and having signed the informed consent

Exclusion Criteria:

* Pregnancy
* Immunodeficiency
* Refuse or unable to sign informed consent
* Chronic disease (i.e. COPD, Crohn, cardiac…)

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2006-08; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
CO2 absorption | measurements for 60 to 240 minutes on average during surgery
  Measurement of end tidal CO2 during laparoscopic surgery; a decrease would improve safety (less hypercarbia)

SECONDARY OUTCOMES:
hemodynamic alterations | measurements for 60 to 240 minutes on average during surgery
  control of other hemodynamic alterions during laparoscopic surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Leuven, campus Gasthuisberg, Leuven, Belgium